CLINICAL TRIAL: NCT06130956
Title: The Effect of a 2-week Preoperative Vegan Diet Versus Omnivorous Diet on the Protein Turnover in the Osteoarthritic Knee
Acronym: KneeT-vegan
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: Gelderse Vallei Hospital (Other); Rijnstate Hospital (Other)
Responsible Party: Principal Investigator, Lisette de Groot, prof.dr.ir., Wageningen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022023
Record Dates: First submitted 2023-11-08; First posted 2023-11-14 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Osteo Arthritis Knee; Protein Synthesis
MeSH Terms: interventions — Diet, Vegan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vegan group (Experimental): Subjects in the vegan group will receive a vegan diet during the 2-week preoperative period.
  Interventions: Dietary Supplement: Vegan diet
- Omnivorous group (Active Comparator): Subjects in the omnivorous group will receive an omnivorous diet during the 2-week preoperative period.
  Interventions: Dietary Supplement: Omnivorous diet

INTERVENTIONS:
Dietary Supplement: Vegan diet — Vegan diet for 2 weeks before surgery
  Arms: Vegan group
Dietary Supplement: Omnivorous diet — Omnivorous diet for 2 weeks before surgery
  Arms: Omnivorous group

SUMMARY:
Rationale: Protein from plant-based foods may be unable to stimulate protein synthesis due to a suboptimal essential amino acid content and a lower digestibility. However, a more optimal amino acid profile may be achieved by increasing portions sizes and blending multiple plant-based sources. Studies investigating the anabolic properties of vegan diets (total elimination of animal-based foods) rather than single plant-based foods in older adults are scarce. It remains unknown if a vegan diet can also affect protein synthesis rates in other musculoskeletal tissues than muscle.

Primary objective: To assess the effects of a 2-week preoperative vegan diet in comparison to an omnivorous diet on protein synthesis rates in Hoffa's fat pad, synovium, tendon, bone, ligaments, menisci, and cartilage in older adults with knee osteoarthritis undergoing total knee arthroplasty.

Secondary objective: To assess the effects of a 2-week preoperative vegan diet in comparison to an omnivorous diet on blood pressure and plasma amino acids in older adults with knee osteoarthritis undergoing total knee arthroplasty.

Study design: Multi-center, randomized, controlled trial with an intervention and a control group.

Study population: 40 older adults (60 - 80 years) with osteoarthritis of the knee undergoing total knee replacement.

Intervention: Controlled vegan diet versus controlled omnivorous diet, for a duration of 14 days.

Main study parameters/endpoints: Primary study parameters are protein synthesis rates of Hoffa's fat pad, synovium, tendon, bone, ligament, menisci, and cartilage. Secondary parameters include blood pressure and plasma amino acids.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent;
* Patients scheduled for total knee arthroplasty;
* BMI between 20-32 kg/m2;
* Aged 60 - 80 years;
* Mentally competent, as judged by the treating physician;

Exclusion Criteria:

* Following a vegetarian or vegan diet or a diet that affects protein intake during the six months prior to the study;
* Participating in a structured progressive exercise training program in the past three months;
* Lost more than 4 kg body weight during three months prior to the study;
* Chronic use of medications that affect protein metabolism (i.e. systemic corticosteroids, or prescription strength acne medications);
* Being diagnosed with one of the following: diabetes mellitus, rheumatoid arthritis, peripheral artery disease Fontaine III or IV, COPD GOLD III or IV, neoadjuvant chemotherapy or radiotherapy, phenylketonuria, collagen disorders (e.g. Marfan and Ehler-Danlos);
* Alcohol abuse;
* Surgical intervention to the knee in the past four weeks;
* Total parenteral nutrition at day of surgery;
* Glomerular filtration rate (GFR) <20 mL/min/1.73 m2;
* Allergic or intolerant to any product included in the diets;
* Osteoarthritis of the knee secondary to septic arthritis, osteonecrosis, fracture, osteochondritis dissecans, or malignant processes;
* Any other medical condition that may interfere with the safety of the participants or the outcome parameters, in the investigators judgement;
* Not willing to stop nutritional supplements, with the exception of vitamin D and supplements on medical advice.
* Investigator's uncertainty about the willingness or ability of the participant to comply with the protocol instructions;
* Participation in other studies that may have an impact on the outcomes during the three months before the start of the current study.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in tissue-specific protein synthesis rates | During the 2-week preoperative period
  Tissue-specific protein synthesis rates in the knee using D2O dosing methodology

SECONDARY OUTCOMES:
Change in blood pressure | Measured at baseline and 1 day before surgery
  Blood pressure measurement using an CE-certified ambulatory blood pressure monitor
Change in plasma amino acids | During the 2-week preoperative period
  Difference in circulating concentrations between the two diets. In addition, it will be investigated if plasma amino acids can be used as a marker for dietary intake.

CONTACTS AND LOCATIONS:
Overall Officials: Lisette de Groot, PhD, Principal Investigator — Wageningen University
Locations (2):
- Netherlands (2):
  - Rijnstate Hospital, Arnhem
  - Hospital Gelderse Vallei, Ede

IPD SHARING:
Plan to Share IPD: No